CLINICAL TRIAL: NCT01079481
Title: A Phase I Study of Combination Anticancer Therapy of Paclitaxel and Everolimus for Relapsed or Refractory Small Cell Lung Cancer
Brief Title: Combination Anticancer Therapy of Paclitaxel and Everolimus for Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-034
Record Dates: First submitted 2010-02-08; First posted 2010-03-03 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Small Cell Lung Cancer
Keywords: Relapsed or Refractory Small Cell Lung Cancer; Paclitaxel; Everolimus
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — Paclitaxel; Everolimus

ARMS (1):
- taxol plus everolimus (Experimental)
  Interventions: Drug: taxol plus everolimus

INTERVENTIONS:
Drug: taxol plus everolimus — taxol 175mg/m2 every 3 weeks plus everolimus every day. The dose of everolimus will be started from 2.5mg per day, and increasing to 5mg per day and to 10mg per day.

SUMMARY:
The objective of this phase I study is to determine the maximum tolerated dose (MTD) of combination therapy of paclitaxel and everolimus in small cell lung cancer patient with previous treatment history.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) accounts for 15% to 20% of all lung cancer, and more than half of these patients are diagnosed with extensive-stage disease (ED). SCLC is a particularly aggressive form of lung cancer with a tendency for rapid tumor growth, early dissemination and high frequency of the metastasis In this study, we evaluate the MTD of everolimus combined with paclitaxel combination chemotherapy in SCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed small cell lung cancer
2. Regarding a limited disease, the disease in a patient, who had concurrent chemoradiation therapy before, is relapsed or progressing, the patient should have received the first line platinum-based anticancer therapy. The disease should be progressing/relapsed during or after the previous treatment.
3. Regarding an extensive disease, the progression/relapse of the disease during or after the first line platinum-based anticancer therapy should be confirmed.
4. Patient with asymptomatic or treated brain metastasis.
5. Patients without current concomitant chemotherapy
6. Patients without current concomitant radiotherapy
7. Patients who are not receiving chronic treatment with steroids or another immunosuppressive agent.
8. Patients with at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST).
9. Patients aged 18 years or older
10. ECOG performance status 0-2
11. Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; hemoglobin > 9g/dL; -; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; creatinine clearance ≥ 50mL/min.
12. Patients who signed and dated the informed consent form prior to specific study procedures.
13. Patients who can comply with the scheduled follow-up and toxicity management procedure.'

Exclusion Criteria:

1. Patients with history of treatment with mTOR inhibitors
2. Pregnant with gastrointestinal problem impairing absorption of drugs
3. Patients who could not use appropriate method of contraception
4. Pregnant or feeding patients
5. Other medically ill patients
6. Severe heart/pulmonary disease
7. DM patients
8. Other malignancy except cured skin cancer or uterine cervix carcinoma in situ
9. High cholesterolemia greater than grade 3
10. Patients with symptomatic brain metastasis
11. Chronic hepatitis or liver cirrhosis (patients with HBsAg positive, IgM anti-HBc positive or HCV Ab positive)
12. Patients receiving immunosuppressant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of everolimus when combined with fixed dose of paclitaxel in small cell lung cancer patients | 18 months

SECONDARY OUTCOMES:
To evaluate the safety when paclitaxel plus everolimus are given to patients with small cell lung cancer | 18 months
To evaluate the objective response rate by RECIST 1.1 criteria | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, M.D., Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea